CLINICAL TRIAL: NCT06552221
Title: Finistere Myeloma Observatory: Retrospective Study of Chromosome 1 Abnormalities and Prognostic Value of a CKS1B (on 1q21)/CDKN2C (on 1p32) Copy Number Ratio in Myeloma.
Brief Title: Finistere Myeloma Observatory (OMYFIN)
Acronym: OMYFIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: OMYFIN (29BRC20.0178)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current molecular risk stratification of multiple myeloma (MM), based on the presence of t(4 ;14) and 17p deletion, cannot fully explain treatment outcome heterogeneity, as other features also predict prognosis. About 30% of genetic events map to chromosome 1 : most upregulated genes to 1q and most downregulated ones to 1p. CKS1B gains on 1q21 and CDKN2C loss on 1p32, both favoring cell cycle progression, portended impaired outcome in many but not all studies. Based on their recurrence and considering their functional convergence, we hypothesized CKS1B/CDKN2C copy number ratio to be a risk factor fitter than each aberration alone.

DETAILED DESCRIPTION:
This single-center retrospective study, is designed to enroll all consecutive newly diagnosed adult patients aged ≥18 years, transplant-eligible and not. All patients are routinely tested for CKS1B and CDKN2C and treated according to consensus guidelines. Data are being collected from 2012. For each subject, we calculate a FISH-based ratio by CKS1B on CDKN2C copy number : it is equal to 1 with no change in copy number and >1 in case of CKS1B gains, CDKN2C loss or both. In patients with CDKN2C biallelic loss, the ratio is not equal to 0, but to CKS1B copy number, as functional consequence should prevail over arithmetic result. We will, then, analyze separately the impact of CKS1B gains, CDKN2C loss and CKS1B/CDKN2C ratio on PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

* Age at or over 18 years
* Symptomatic multiple myeloma
* Informed consent given
* FISH-based cytogenetic results obtained

Exclusion Criteria:

* Age under 18 years
* MGUS or SMM
* No informed consent
* No FISH-based cytogenetic results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive symptomatic multiple myeloma patients seen and treated i Hematology Department at Brest University Hospital from January 1, 2012 whose CKS1B/CDKN2C copy number ratio at diagnosis is calculable.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Response rate | 10 years
  The aim is to assess the impact of CKS1B/CDKN2C copy number ratio on response rate

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 10 years
  The aim is to assess the impact of CKS1B/CDKN2C copy number ratio on PFS

OTHER OUTCOMES:
Overall survival (OS) | 10 years
  The aim is to assess the impact of CKS1B/CDKN2C copy number ratio on OS

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Richard Eveillard, MD, Principal Investigator — CHU de Brest
Locations (1):
- CHRU de Brest, Brest, France